CLINICAL TRIAL: NCT07096336
Title: Effect of Vitamin D3 Supplementation on Brain Waves in Male Parkinson's Disease Patients With Hypovitaminosis D : A Quantitative Electroencephalogram Analysis
Brief Title: Effect of Vitamin D3 on Brain Waves in Male Parkinson's Patients With Low Vitamin D: A qEEG Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Jannatul Ferdoush Sumi, MD resident , Department of Physiology, Bangladesh Medical University, Principal investigator,, Bangladesh Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5586
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Parkinson's disease; Vitamin D3; Quantitative EEG (qEEG); Brain wave; 25-hydroxyvitamin D; Spectral power; Dopaminergic neurons; EEG frequency bands; Neurodegeneration
MeSH Terms: conditions — Parkinson Disease; Nerve Degeneration | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Experimental study ( Interventional self controlled experimental trial) where 15 participants will be enrolled to compare their baseline data with post interventional data
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Male Parkinson's disease patients with hypovitaminosis D (Experimental): 15 Male Parkinson's disease patients with hypovitaminosis D will be supplemented with vitamin D orally 50,000 IU/week for 8 weeks
  Interventions: Dietary Supplement: vitamin D3 capsule

INTERVENTIONS:
Dietary Supplement: vitamin D3 capsule — Administration of vitamin D3 capsule 50,000 IU/week for 8 weeks

SUMMARY:
This is an experimental study (Interventional self-controlled trial, pretest-posttest design). The goal of this clinical trial is to evaluate the effect of vitamin D3 supplementation on quantitative EEG in male Parkinson's disease patients with hypovitaminosis D.

The main question it aims to answer is:

Vitamin D3 supplementation has effect on brain waves in male Parkinson's disease patients with hypovitaminosis D.

Researcher will compare the effect of vitamin D3 supplementation on brain waves in male Parkinson's disease patients with hypovitaminosis D with their pre intervention ( baseline ) condition on brain waves to assess whether there will be any improvement of brain electrical activity by quantitative electroencephalogram (QEEG).

Participants will :

Take vitamin D3 orally for 8 weeks (50,000 IU/week) Visit the medical university after 8 weeks for evaluation of serum 25(OH)D level and QEEG Must bring the empty strips of vitamin D supplement with them during their visit.

DETAILED DESCRIPTION:
This self-controlled experimental study will be conducted at the Department of Physiology, BMU, Dhaka, between March 2025 and February 2026. Fifteen male patients with Parkinson's disease (PD) and confirmed hypovitaminosis D will be recruited from the Neurology Outpatient Department. Each participant will undergo serum 25(OH)D level assessment and baseline EEG recording (Session A1). Following this, they will receive vitamin D3 supplementation orally (50,000 IU weekly) for 8 weeks. After the intervention period, serum 25-hydroxyvitamin D level will be reassessed and EEG recording will be done again (Session AD). The EEG data will be collected using an EEG Traveler BrainTech 32+ CMEEG-01 device using Fast Fourier Transform (FFT) to derive spectral parameters including absolute power, relative power, peak power frequency (PPF), median power frequency (MPF), and spectral edge frequency (SEF) across delta, theta, alpha, and beta frequency bands. Statistical analysis will be performed using SPSS version 25. Data will be tested for normality using the Shapiro-Wilk test. Paired t-tests or Wilcoxon signed-rank tests will be applied for within-group comparisons, with statistical significance set at p ≤ 0.05.

This research aims to fill this gap by using quantitative EEG to investigate if vitamin D3 supplementation modulates brain electrical activity in PD patients who are deficient or insufficient in vitamin D. The findings could contribute to a better understanding of the neurophysiological effects of vitamin D3 and support its potential as an adjunctive therapeutic strategy in managing PD.

ELIGIBILITY:
Inclusion Criteria:

* Male Patients with PD up to stage 3 according to Hoehn and Yahr (H-Y) scale
* Age: 51years to70 years
* BMI: 18.5-24.9 kg/m2
* Hypovitaminosis D (Serum 25(OH)D level <30 ng/ml)
* Patients on Levodopa therapy

Exclusion Criteria:

* Already taking vitamin D3 supplements
* Current use of medication/substances known to affect neuronal excitability or EEG patterns, such as - sedatives, antidepressant, antipsychotics, alcohol.
* Patients who are currently suffering from following diseases

  * Neurological disorders (Migraine, epilepsy)
  * Cardiovascular disorders (Myocardial infarction, hypertension, cardiac arrhythmia, heart failure)
  * Respiratory disorders (Bronchial asthma, COPD)
  * Psychiatric illness (e.g., schizophrenia, major depression, bipolar disorder, severe dementia)
* With biochemical evidence of-

  * Hypercalcemia
  * Renal insufficiency
  * Liver diseases
  * Endocrine disorders (uncontrolled diabetes mellitus, Hypothyroidism, Hyperthyroidism)
* Active smoker

Ages: 51 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in absolute power in alpha, beta, theta, and delta frequency bands from baseline to 8 weeks | 8 weeks
  Measured using FFT-based quantitative EEG (qEEG) analysis. Unit of Measure: microvolts squared (µV²)
Change in relative power in alpha, beta, theta, and delta frequency bands from baseline to 8 weeks | 8 weeks
  Measured using FFT-based quantitative EEG (qEEG) analysis. Unit of Measure: percentage (%)
Change in peak power frequency in alpha, beta, theta, and delta bands from baseline to 8 weeks | 8 weeks
  Measured from global EEG spectrum using FFT-based qEEG analysis. Unit of Measure: Hertz (Hz)
Change in median power frequency from baseline to 8 weeks | 8 weeks
  Measured from global EEG spectrum using FFT-based qEEG analysis. Unit of Measure: Hertz (Hz)
Change in spectral edge frequency (SEF 90) from baseline to 8 weeks | 8 weeks
  Calculated from global EEG spectrum using FFT-based qEEG analysis. Unit of Measure: Hertz (Hz)

CONTACTS AND LOCATIONS:
Locations (1):
- Bangladesh medical university, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No